CLINICAL TRIAL: NCT01913028
Title: A Phase 1, Single Centre, Single-blind, Randomized, Placebo-controlled Parallel-group Study to Evaluate the Safety, Tolerability, Pharmacokinetics and Immunogenicity of MEDI9929 After Administration of Single Ascending Doses in Healthy Male Japanese Subjects
Brief Title: A Phase 1 Study to Evaluate the Safety, Tolerability, Pharmacokinetics and Immunogenicity of MEDI9929 After Single Administration in Healthy Male Japanese Subjects
Status: Completed | Phase: Phase 1 | Type: Interventional
Sponsor: AstraZeneca (Industry)
Collaborators: MedImmune LLC (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Basic Science
Other Study IDs: D5180C00003
Record Dates: First submitted 2013-07-30; First posted 2013-07-31 (Estimated); Last update posted 2014-02-12 (Estimated); Status verified 2014-02

CONDITIONS: Healthy
Keywords: safety, tolerability, pharmacokinetics,immunogenicity, MEDI9929, Japanese
MeSH Terms: interventions — tezepelumab

STUDY DESIGN:
Who Masked: Participant
Oversight: Data Monitoring Committee: No

ARMS (2):
- MEDI9929 (Experimental): Solution of MEDI9929, SC
  Interventions: Drug: MEDI9929
- Placebo (Placebo Comparator): Placebo solution for MEDI9929, SC
  Interventions: Drug: Placebo

INTERVENTIONS:
Drug: MEDI9929 — 1st cohort : Dose 1 MEDI9929 or placebo 2nd cohort : Dose 2 MEDI9929 or placebo 3rd cohort : Dose 3 MEDI9929 or placebo
  Arms: MEDI9929
Drug: Placebo — 1st cohort : Dose 1 MEDI9929 or placebo 2nd cohort : Dose 2 MEDI9929 or placebo 3rd cohort : Dose 3 MEDI9929 or placebo
  Arms: Placebo

SUMMARY:
The purpose of this study is to assess safety, tolerability, pharmacokinetics and immunogenicity of MEDI9929 following administration of single ascending doses in healthy male Japanese subjects.

DETAILED DESCRIPTION:
This is a Phase I, single centre, randomised, single-blind, placebo-controlled, single ascending dose parallel study in healthy male Japanese subjects. Up to 3 dose levels of MEDI9929 will be investigated.

Primary object is to assess the safety and tolerability of single ascending subcutaneous (SC) doses of MEDI9929 in healthy male Japanese subjects. Secondary objectives are to characterize the pharmacokinetics (PK) of MEDI9929 in healthy male Japanese subjects and to evaluate the immunogenicity (IM) of MEDI9929 in healthy male Japanese subjects.

Up to 24 healthy subjects aged 20 to 45 years will participate in a maximum of 3 cohorts.

Eight subjects will participate in each cohort. Subjects will be randomized in a 3:1 ratio (active: placebo) and will receive a single dose of either MEDI9929 or placebo. Each subject will only participate in one cohort.

The first cohort will receive Dose 1 MEDI9929 (n=6) or placebo (n=2), the second cohort will receive Dose 2 MEDI9929 (n=6) or placebo (n=2), and the third cohort will receive Dose 3 MEDI9929 (n=6) or placebo (n=2).

Following a screening period of a maximum of 28 days, subjects will stay at the study facility for eight nights starting from the day before dosing (Day -1) to Day 8. The follow up period after the dosing will be 84 days (112 days for cohort 3). Subjects will receive a single dose of MEDI9929 or placebo subcutaneously on Day 1 and safety monitoring and serial collection of blood samples for PK evaluation will be followed throughout the study period.

ELIGIBILITY:
Inclusion Criteria:

1. Provision of signed and dated, written informed consent prior to any study specific procedures.
2. Healthy Japanese male subjects aged 20 - 45 years age with a body mass index(BMI) between 18 - 27 kg/m2 at the time of screening
3. Sterilized males must be at least 1-year post vasectomy or non-sterilized males who are sexually active with a female partner of childbearing potential must use a highly effective method of contraception from Day 1 through Day 85 (through Day 113 for cohort 3); It is highly recommended for both partners to use contraception, preferably one hormonal or intrauterine device (females) and one barrier method (males).

   Were men who agree to use birth control for 4 months after the last dose of investigational product and to not donate sperm for 4 months after the last dose of investigational product
4. Able to comply with the requirements of the protocol

Exclusion Criteria:

1. Had history or evidence of a clinically significant disorder, condition, or disease (including cardiopulmonary, oncologic, immunologic, autoimmune, collagen vascular, renal, metabolic, hematologic, or psychiatric), that in the opinion of the investigator, would pose a risk to subject safety or interfere with the study evaluation, procedures, or completion
2. Any acute illness in the 14 days before Day 1
3. Had evidence of any active or suspected bacterial, viral, fungal, or parasitic infections within the past 30 days before randomization (eg, common cold, viral syndrome, flu-like symptoms), or a high risk, in the opinion of the investigator, for parasitic disease
4. Clinically relevant abnormalities in physical examinations, vital signs, clinical chemistry, hematology or urinalysis as judged by the investigator
5. Has a history of anaphylaxis to another therapeutic monoclonal antibody or biologic therapy

Ages: 20 Years to 45 Years | Sex: Male | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 64 (Actual)
Dates: Start 2013-08; Primary Completion 2014-01 (Actual); Study Completion 2014-01 (Actual)

PRIMARY OUTCOMES:
Description of the Safety and tolerability profile of MEDI9929 | 84 days for cohort 1/2, 112 days for cohort 3
  To investigate the safety and tolerability (Adverse events, blood pressure and pulse, Electrocardiogram, Body temperature, respiratory rate, Haematology, Clinical Chemistry, Urinalysis, and physical examination) of MEDI9929 following administration of single ascending doses.

SECONDARY OUTCOMES:
Description of Pharmacokinetics profile for MEDI9929 | 84 days for cohort 1/2, 112 days for cohort 3
  To characterize the pharmacokinetics of MEDI9929 after single SC dose in healthy male Japanese subjects. Where possible, the following PK parameters will be determined: Apparent SC clearance [CL/F], apparent SC volume of distribution [Vz/F], maximum observed serum concentration, [Cmax], time at which maximum concentration is observed [tmax], area under the serum concentration time curve from time zero to infinity [AUC0-inf] and to last observation [AUC(0-t)], elimination half-life [t½, z]
Description of Immunogenicity profile for MEDI9929 | 84 days for cohort 1/2, 112 days for cohort 3
  Description of immunogenicity in terms of positive or negative for the presence of antidrug antibodies against MEDI9929 in blood.

CONTACTS AND LOCATIONS:
Overall Officials: Kei Sakamoto, MD, PhD, Principal Investigator — Kyushu Clinical Pharmacology Research Clinic, Medical Co. LTA
Locations (2):
- Japan (2):
  - Kyushu Clinical Pharmacology Research Clinic, Medical Co. LTA, Fukuoka, Hakata
  - Research Site, Fukuoka